CLINICAL TRIAL: NCT07119658
Title: Targeting Metabolic Syndrome From the Emergency Department Through Mixed-Methods: Pilot Trial
Acronym: METS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Society for Academic Emergency Medicine (Other)
Responsible Party: Principal Investigator, Lauren Stewart, Assistant Professor of Emergency Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25821; RE2022-0000000327 (Other Grant/Funding Number: Society for Academic Emergency Medicine Foundation)
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Hyperglycemia; Dyslipidemia; Metabolic Syndrome; Obesity &Amp; Overweight; Diabetes; Hyperlipidemia; Emergency Medicine
Keywords: Metabolic Syndrome; Emergency Department
MeSH Terms: conditions — Hypertension; Hyperglycemia; Dyslipidemias; Metabolic Syndrome; Obesity; Overweight; Diabetes Mellitus; Hyperlipidemias; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The composite intervention will include an educational video outlining the adverse effects of metabolic syndrome and the benefit of walking (which patients will watch at time of enrollment in the emergency department), a written exercise "prescription" with a defined goal of walking 150 minutes per week, a Fitbit accelerometer device to track activity, resources for healthy eating practices, periodic text message reminders over the 3 month study period, and an urgent referral to primary care and our health system's Healthy Me clinic for follow-up visit.
  Interventions: Behavioral: Composite intervention to address MetS
- Control (No Intervention): The control group will receive usual care upon discharge from the emergency department. They will be given a Fitbit accelerometer device to wear for the study period to serve as a comparison but will not receive any specific recommendations for active or any additional component of the composite intervention.

INTERVENTIONS:
Behavioral: Composite intervention to address MetS — The composite intervention includes six components: 1. All patients will be provided a Fitbit Charge device at ED discharge with instructions to wear on their wrist for study duration. 2. Participants in the intervention group will first watch a brief (~5 minute) educational video outlining the adverse effects of MetS and the benefit of walking, via iPad tablet. 3. Participants in the intervention group will also be given accompanying written "exercise prescription" encouraging them to walk 150 minutes per week. 4. Reminder texts encouraging continued walking behavior (i.e. "Remember to get in your steps!") will be sent to the intervention group, at approximate 2-3x/week intervals for the 3-month follow-up period. 5. The intervention group will also be provided written resources for healthy eating practices upon ED discharge. 6. All intervention group participants will receive referrals into primary care clinic and the Eskenazi Health "Healthy Me" Program for follow-up.
  Arms: Intervention

SUMMARY:
The objective of this study is to pilot a multifaceted, optimized intervention for metabolic syndrome (MetS) in emergency department patients to establish feasibility. Participants (n=20) will be randomized to intervention or control (usual care). The composite intervention will include an educational video outlining the adverse effects of MetS and the benefit of walking, a written exercise prescription with a defined goal of walking 150 minutes per week, a Fitbit accelerometer device, resources for healthy eating practices, periodic text message reminders, and an urgent referral to primary care and our health system's Healthy Me clinic for follow-up visit. Investigators hypothesize that this approach will change patient understanding and motivation to increase physical activity and healthy eating habits.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adults (18 years of age) presenting to the emergency department setting
* BMI 30 kg/m2
* Prior diagnosis of at least one additional comorbid component of metabolic syndrome: hypertension, hyperglycemia, dyslipidemia
* Clinical plan for discharge

Exclusion Criteria:

* Age <18 years
* Pregnant patients
* Unable to safely ambulate (including patient or family perception of inability to safely ambulate)
* Lack of access to smart phone
* Unable or unwilling to wear Fitbit accelerometer device
* Unable to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mean daily steps | From enrollment to the end of the 3 month study period
  Investigators will collect activity data utilizing a Fitbit accelerometer device. The primary outcome will be the mean number of daily steps averaged from 3 months of monitoring, compared between groups.

SECONDARY OUTCOMES:
Minutes of moderate to vigorous physical activity | From enrollment to the end of the 3 month study period
  Investigators will collect activity data utilizing a Fitbit accelerometer device. As a secondary outcome, investigators will measure and compare minutes of moderate to vigorous physical activity (MVPA), as this metric will incorporate intensity of activity.
Psychometric survey: the Dietary Screener Questionnaire | At enrollment and 3 month follow-up
  Participants will complete the Dietary Screener Questionnaire survey at baseline and 3-months.
Psychometric surveys: International Physical Activity Questionnaire | At enrollment and 3 month follow-up
  Participants will complete the International Physical Activity Questionnaire survey at baseline and 3-months. This is reported on a continuous scale as physical activity metabolic equivalent of task (MET)-min per day or week.
Psychometric surveys: PROMIS General Life Satisfaction -- Short Form 5a | At enrollment and 3 month follow-up
  Participants will complete the NIH PROMIS General Life Satisfaction -- Short Form 5a survey at baseline and 3-months. (min value: 5, max value: 35, higher score = higher life satisfaction)
Psychometric surveys: PROMIS Physical Function -- Short Form 4a | At enrollment and 3 month follow-up
  Participants will complete the NIH PROMIS Physical Function -- Short Form 4a survey at baseline and 3-months. (min value: 4, max value: 20, higher score = higher physical functioning)
Psychometric surveys: PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Daily Activities -- Short Form 8a | At enrollment and 3 month follow-up
  Participants will complete the NIH PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Daily Activities -- Short Form 8a survey at baseline and 3-months. (min value: 8, max value: 40, higher score = higher self-efficacy)
Number of participants with a repeat visit to the emergency department | From enrollment to 3 month follow-up
  Investigators will assess ED recidivism over the 3-month follow-up period, which will be defined as any repeat visit to the emergency department over the study period. This will be assessed primarily through review of the electronic medical record for any new ED encounter that occurred after initial enrollment date.

OTHER OUTCOMES:
Successful linkage into outpatient clinic follow-up | From enrollment to 3 month follow-up
  Investigators will determine whether intervention patients were able to successfully follow up in the health system's outpatient clinic with the referral provided. This will be determined through review of the electronic medical record.
Number of days wearing the Fitbit accelerometer during study period | From enrollment to 3 month follow-up
  Investigators will describe the number of totals days participants actually wore the Fitbit accelerometer device over the study period, allowing for activity data collection.
Demographic data | This will be collected on Day 1 (i.e. day of screening and approaching for enrollment)
  As an additional exploration, we will collect pertinent data on the screening and enrollment process, including demographic data on which patients are screened, approached, and ultimately enrolled. We will ask those who decline enrollment to briefly provide us information (i.e. short-form, open-ended response) on why they are declining to participate, to gain further knowledge on the targeted ED population for this intervention.
Semi-structured interview data | At 3-month follow-up (for those in intervention group)
  To better understand reasons for failure and success of adherence to the composite intervention, we will also conduct semi-structured interviews at three-month follow-up of patients in the intervention group. Thematic analysis will be performed to identify theoretical constructs, processes, and themes surrounding the patients' experience with the composite intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney & Lois Eskenazi Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sista AK, Klok FA. Late outcomes of pulmonary embolism: The post-PE syndrome. Thromb Res. 2018 Apr;164:157-162. doi: 10.1016/j.thromres.2017.06.017. Epub 2017 Jun 16. PMID 28641836
- [Background] Piercy KL, Troiano RP, Ballard RM, Carlson SA, Fulton JE, Galuska DA, George SM, Olson RD. The Physical Activity Guidelines for Americans. JAMA. 2018 Nov 20;320(19):2020-2028. doi: 10.1001/jama.2018.14854. PMID 30418471
- [Background] Lee IM, Shiroma EJ, Kamada M, Bassett DR, Matthews CE, Buring JE. Association of Step Volume and Intensity With All-Cause Mortality in Older Women. JAMA Intern Med. 2019 Aug 1;179(8):1105-1112. doi: 10.1001/jamainternmed.2019.0899. PMID 31141585
- [Background] Dontje ML, de Groot M, Lengton RR, van der Schans CP, Krijnen WP. Measuring steps with the Fitbit activity tracker: an inter-device reliability study. J Med Eng Technol. 2015;39(5):286-90. doi: 10.3109/03091902.2015.1050125. Epub 2015 May 27. PMID 26017748
- [Background] Feehan LM, Geldman J, Sayre EC, Park C, Ezzat AM, Yoo JY, Hamilton CB, Li LC. Accuracy of Fitbit Devices: Systematic Review and Narrative Syntheses of Quantitative Data. JMIR Mhealth Uhealth. 2018 Aug 9;6(8):e10527. doi: 10.2196/10527. PMID 30093371
- [Background] Stich C, Knauper B, Tint A. A scenario-based dieting self-efficacy scale: the DIET-SE. Assessment. 2009 Mar;16(1):16-30. doi: 10.1177/1073191108322000. Epub 2008 Aug 14. PMID 18703821
- [Background] McAuley E. Self-efficacy and the maintenance of exercise participation in older adults. J Behav Med. 1993 Feb;16(1):103-13. doi: 10.1007/BF00844757. PMID 8433355
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Mattila J, Ding H, Mattila E, Sarela A. Mobile tools for home-based cardiac rehabilitation based on heart rate and movement activity analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:6448-52. doi: 10.1109/IEMBS.2009.5333540. PMID 19964430
- [Background] Brouwers RW, Kraal JJ, Traa SC, Spee RF, Oostveen LM, Kemps HM. Effects of cardiac telerehabilitation in patients with coronary artery disease using a personalised patient-centred web application: protocol for the SmartCare-CAD randomised controlled trial. BMC Cardiovasc Disord. 2017 Jan 31;17(1):46. doi: 10.1186/s12872-017-0477-6. PMID 28143388
- [Background] Satia JA. Diet-related disparities: understanding the problem and accelerating solutions. J Am Diet Assoc. 2009 Apr;109(4):610-5. doi: 10.1016/j.jada.2008.12.019. No abstract available. PMID 19328255
- [Background] Siopis G, Chey T, Allman-Farinelli M. A systematic review and meta-analysis of interventions for weight management using text messaging. J Hum Nutr Diet. 2015 Feb;28 Suppl 2:1-15. doi: 10.1111/jhn.12207. Epub 2014 Jan 31. PMID 24480032
- [Background] Smith DM, Duque L, Huffman JC, Healy BC, Celano CM. Text Message Interventions for Physical Activity: A Systematic Review and Meta-Analysis. Am J Prev Med. 2020 Jan;58(1):142-151. doi: 10.1016/j.amepre.2019.08.014. Epub 2019 Nov 21. PMID 31759805
- [Background] Fox SM 3rd, Naughton JP, Haskell WL. Physical activity and the prevention of coronary heart disease. Ann Clin Res. 1971 Dec;3(6):404-32. No abstract available. PMID 4945367
- [Background] KARVONEN MJ, KENTALA E, MUSTALA O. The effects of training on heart rate; a longitudinal study. Ann Med Exp Biol Fenn. 1957;35(3):307-15. No abstract available. PMID 13470504
- [Background] Yoong SL, Hall A, Stacey F, Grady A, Sutherland R, Wyse R, Anderson A, Nathan N, Wolfenden L. Nudge strategies to improve healthcare providers' implementation of evidence-based guidelines, policies and practices: a systematic review of trials included within Cochrane systematic reviews. Implement Sci. 2020 Jul 1;15(1):50. doi: 10.1186/s13012-020-01011-0. PMID 32611354
- [Background] Onken LS, Carroll KM, Shoham V, Cuthbert BN, Riddle M. Reenvisioning Clinical Science: Unifying the Discipline to Improve the Public Health. Clin Psychol Sci. 2014 Jan 1;2(1):22-34. doi: 10.1177/2167702613497932. PMID 25821658
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Stewart LK, Sarmiento EJ, Kline JA. Statin Use is Associated with Reduced Risk of Recurrence in Patients with Venous Thromboembolism. Am J Med. 2020 Aug;133(8):930-935.e8. doi: 10.1016/j.amjmed.2019.12.032. Epub 2020 Mar 12. PMID 32171773
- [Background] Stewart LK, Beam DM, Casciani T, Cameron SJ, Kline JA. Effect of metabolic syndrome on mean pulmonary arterial pressures in patients with acute pulmonary embolism treated with catheter-directed thrombolysis. Int J Cardiol. 2020 Mar 1;302:138-142. doi: 10.1016/j.ijcard.2019.12.043. Epub 2019 Dec 26. PMID 31948673
- [Background] Stewart LK, Nordenholz KE, Courtney M, Kabrhel C, Jones AE, Rondina MT, Diercks DB, Klinger JR, Kline JA. Comparison of acute and convalescent biomarkers of inflammation in patients with acute pulmonary embolism treated with systemic fibrinolysis vs. placebo. Blood Coagul Fibrinolysis. 2017 Dec;28(8):675-680. doi: 10.1097/MBC.0000000000000669. PMID 28957940
- [Background] Vaughn LM, Nabors L, Pelley TJ, Hampton RR, Jacquez F, Mahabee-Gittens EM. Obesity screening in the pediatric emergency department. Pediatr Emerg Care. 2012 Jun;28(6):548-52. doi: 10.1097/PEC.0b013e318258ada0. PMID 22653451
- [Background] Prendergast HM, Close M, Jones B, Furtado N, Bunney EB, Mackey M, Marquez D, Edison M. On the frontline: pediatric obesity in the emergency department. J Natl Med Assoc. 2011 Sep-Oct;103(9-10):922-5. doi: 10.1016/s0027-9684(15)30448-x. PMID 22364061
- [Background] Haber JJ, Atti S, Gerber LM, Waseem M. Promoting an obesity education program among minority patients in a single urban pediatric Emergency Department (ED). Int J Emerg Med. 2015 Dec;8(1):38. doi: 10.1186/s12245-015-0086-z. Epub 2015 Oct 28. PMID 26511854
- [Background] Milne F, Leech-Porter K, Atkinson P, Lewis D, Fraser J, Hull S. Combatting Sedentary Lifestyles: Can Exercise Prescription in the Emergency Department Lead to Behavioral Change in Patients? Cureus. 2020 Feb 21;12(2):e7071. doi: 10.7759/cureus.7071. PMID 32226672
- [Background] Peiris CL, Taylor NF, Hull S, Anderson A, Belski R, Fourlanos S, Shields N. A Group Lifestyle Intervention Program Is Associated with Reduced Emergency Department Presentations for People with Metabolic Syndrome: A Retrospective Case-Control Study. Metab Syndr Relat Disord. 2018 Mar;16(2):110-116. doi: 10.1089/met.2017.0127. Epub 2018 Jan 23. PMID 29360416
- [Background] Hobbs N, Godfrey A, Lara J, Errington L, Meyer TD, Rochester L, White M, Mathers JC, Sniehotta FF. Are behavioral interventions effective in increasing physical activity at 12 to 36 months in adults aged 55 to 70 years? A systematic review and meta-analysis. BMC Med. 2013 Mar 19;11:75. doi: 10.1186/1741-7015-11-75. PMID 23506544
- [Background] Orrow G, Kinmonth AL, Sanderson S, Sutton S. Effectiveness of physical activity promotion based in primary care: systematic review and meta-analysis of randomised controlled trials. BMJ. 2012 Mar 26;344:e1389. doi: 10.1136/bmj.e1389. PMID 22451477
- [Background] Armitage LC, Whelan ME, Watkinson PJ, Farmer AJ. Screening for hypertension using emergency department blood pressure measurements can identify patients with undiagnosed hypertension: A systematic review with meta-analysis. J Clin Hypertens (Greenwich). 2019 Sep;21(9):1415-1425. doi: 10.1111/jch.13643. Epub 2019 Aug 6. PMID 31385426
- [Background] Chernow SM, Iserson KV, Criss E. Use of the emergency department for hypertension screening: a prospective study. Ann Emerg Med. 1987 Feb;16(2):180-2. doi: 10.1016/s0196-0644(87)80012-4. PMID 3800093
- [Background] Moss R, Craige EK, Levine B, Mittal M, Ahn S, Appold B, Richman M. Influence of Framing: Recruitment to a Diabetes Disease Management Program From an Emergency Department Improves Enrollment and Outcomes. Cureus. 2021 Mar 25;13(3):e14116. doi: 10.7759/cureus.14116. PMID 33907649
- [Background] Bock BC, Becker BM, Niaura RS, Partridge R, Fava JL, Trask P. Smoking cessation among patients in an emergency chest pain observation unit: outcomes of the Chest Pain Smoking Study (CPSS). Nicotine Tob Res. 2008 Oct;10(10):1523-31. doi: 10.1080/14622200802326343. PMID 18946771
- [Background] Boudreaux ED, Moon S, Baumann BM, Camargo CA Jr, O'Hea E, Ziedonis DM. Intentions to quit smoking: causal attribution, perceived illness severity, and event-related fear during an acute health event. Ann Behav Med. 2010 Dec;40(3):350-5. doi: 10.1007/s12160-010-9227-z. PMID 20827518
- [Background] Jiang LG, Zhang Y, Greca E, Bodnar D, Gogia K, Wang Y, Peretz P, Steel PAD. Emergency Department Patient Navigator Program Demonstrates Reduction in Emergency Department Return Visits and Increase in Follow-up Appointment Adherence. Am J Emerg Med. 2022 Mar;53:173-179. doi: 10.1016/j.ajem.2022.01.009. Epub 2022 Jan 12. PMID 35065524
- [Background] Peart A, Lewis V, Brown T, Russell G. Patient navigators facilitating access to primary care: a scoping review. BMJ Open. 2018 Mar 17;8(3):e019252. doi: 10.1136/bmjopen-2017-019252. PMID 29550777
- [Background] Choo EK, Ranney ML, Aggarwal N, Boudreaux ED. A systematic review of emergency department technology-based behavioral health interventions. Acad Emerg Med. 2012 Mar;19(3):318-28. doi: 10.1111/j.1553-2712.2012.01299.x. PMID 22435865
- [Background] Ranney ML, Suffoletto B. Extending our reach: use of mHealth to support patients after emergency care. Ann Emerg Med. 2014 Jun;63(6):755-6. doi: 10.1016/j.annemergmed.2014.01.015. Epub 2014 Jan 31. No abstract available. PMID 24486096
- [Background] Watson DP, Brucker K, McGuire A, Snow-Hill NL, Xu H, Cohen A, Campbell M, Robison L, Sightes E, Buhner R, O'Donnell D, Kline JA. Replication of an emergency department-based recovery coaching intervention and pilot testing of pragmatic trial protocols within the context of Indiana's Opioid State Targeted Response plan. J Subst Abuse Treat. 2020 Jan;108:88-94. doi: 10.1016/j.jsat.2019.06.002. Epub 2019 Jun 6. PMID 31200985
- [Background] Watson DP, Weathers T, McGuire A, Cohen A, Huynh P, Bowes C, O'Donnell D, Brucker K, Gupta S. Evaluation of an emergency department-based opioid overdose survivor intervention: Difference-in-difference analysis of electronic health record data to assess key outcomes. Drug Alcohol Depend. 2021 Apr 1;221:108595. doi: 10.1016/j.drugalcdep.2021.108595. Epub 2021 Feb 15. PMID 33610095
- [Background] D'Onofrio G, Fiellin DA, Pantalon MV, Chawarski MC, Owens PH, Degutis LC, Busch SH, Bernstein SL, O'Connor PG. A brief intervention reduces hazardous and harmful drinking in emergency department patients. Ann Emerg Med. 2012 Aug;60(2):181-92. doi: 10.1016/j.annemergmed.2012.02.006. Epub 2012 Mar 28. PMID 22459448
- [Background] Bernstein SL, Bijur P, Cooperman N, Jearld S, Arnsten JH, Moadel A, Gallagher EJ. A randomized trial of a multicomponent cessation strategy for emergency department smokers. Acad Emerg Med. 2011 Jun;18(6):575-83. doi: 10.1111/j.1553-2712.2011.01097.x. PMID 21676054
- [Background] Adams EJ, Morris L, Marshall G, Coffey F, Miller PD, Blake H. Effectiveness and implementation of interventions for health promotion in urgent and emergency care settings: an umbrella review. BMC Emerg Med. 2023 Apr 6;23(1):41. doi: 10.1186/s12873-023-00798-7. PMID 37024777
- [Background] McKay MP, Vaca FE, Field C, Rhodes K. Public health in the emergency department: overcoming barriers to implementation and dissemination. Acad Emerg Med. 2009 Nov;16(11):1132-7. doi: 10.1111/j.1553-2712.2009.00547.x. PMID 20053233
- [Background] Goldstein LB, Bushnell CD, Adams RJ, Appel LJ, Braun LT, Chaturvedi S, Creager MA, Culebras A, Eckel RH, Hart RG, Hinchey JA, Howard VJ, Jauch EC, Levine SR, Meschia JF, Moore WS, Nixon JV, Pearson TA; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Epidemiology and Prevention; Council for High Blood Pressure Research,; Council on Peripheral Vascular Disease, and Interdisciplinary Council on Quality of Care and Outcomes Research. Guidelines for the primary prevention of stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2011 Feb;42(2):517-84. doi: 10.1161/STR.0b013e3181fcb238. Epub 2010 Dec 2. PMID 21127304
- [Background] Mitka M. Lifestyle changes key to cut stroke risk: guidelines place emergency physicians on front line. JAMA. 2011 Feb 9;305(6):551-2. doi: 10.1001/jama.2011.93. No abstract available. PMID 21304074
- [Background] Marcus BH, Selby VC, Niaura RS, Rossi JS. Self-efficacy and the stages of exercise behavior change. Res Q Exerc Sport. 1992 Mar;63(1):60-6. doi: 10.1080/02701367.1992.10607557. PMID 1574662
- [Background] Young MD, Plotnikoff RC, Collins CE, Callister R, Morgan PJ. A Test of Social Cognitive Theory to Explain Men's Physical Activity During a Gender-Tailored Weight Loss Program. Am J Mens Health. 2016 Nov;10(6):NP176-NP187. doi: 10.1177/1557988315600063. Epub 2015 Aug 14. PMID 26275722
- [Background] Blackwell DL, Clarke TC. State Variation in Meeting the 2008 Federal Guidelines for Both Aerobic and Muscle-strengthening Activities Through Leisure-time Physical Activity Among Adults Aged 18-64: United States, 2010-2015. Natl Health Stat Report. 2018 Jun;(112):1-22. PMID 30248007
- [Background] Wewege MA, Thom JM, Rye KA, Parmenter BJ. Aerobic, resistance or combined training: A systematic review and meta-analysis of exercise to reduce cardiovascular risk in adults with metabolic syndrome. Atherosclerosis. 2018 Jul;274:162-171. doi: 10.1016/j.atherosclerosis.2018.05.002. Epub 2018 May 3. PMID 29783064
- [Background] Ostman C, Smart NA, Morcos D, Duller A, Ridley W, Jewiss D. The effect of exercise training on clinical outcomes in patients with the metabolic syndrome: a systematic review and meta-analysis. Cardiovasc Diabetol. 2017 Aug 30;16(1):110. doi: 10.1186/s12933-017-0590-y. PMID 28854979
- [Background] Stefani L, Galanti G. Physical Exercise Prescription in Metabolic Chronic Disease. Adv Exp Med Biol. 2017;1005:123-141. doi: 10.1007/978-981-10-5717-5_6. PMID 28916931
- [Background] Roberts CK, Hevener AL, Barnard RJ. Metabolic syndrome and insulin resistance: underlying causes and modification by exercise training. Compr Physiol. 2013 Jan;3(1):1-58. doi: 10.1002/cphy.c110062. PMID 23720280
- [Background] McGuire S. Scientific Report of the 2015 Dietary Guidelines Advisory Committee. Washington, DC: US Departments of Agriculture and Health and Human Services, 2015. Adv Nutr. 2016 Jan 15;7(1):202-4. doi: 10.3945/an.115.011684. Print 2016 Jan. No abstract available. PMID 26773024
- [Background] Mozaffarian D. Dietary and Policy Priorities for Cardiovascular Disease, Diabetes, and Obesity: A Comprehensive Review. Circulation. 2016 Jan 12;133(2):187-225. doi: 10.1161/CIRCULATIONAHA.115.018585. PMID 26746178
- [Background] Castro-Barquero S, Ruiz-Leon AM, Sierra-Perez M, Estruch R, Casas R. Dietary Strategies for Metabolic Syndrome: A Comprehensive Review. Nutrients. 2020 Sep 29;12(10):2983. doi: 10.3390/nu12102983. PMID 33003472
- [Background] Parker BK, Manning S, Winters ME. The Crashing Obese Patient. West J Emerg Med. 2019 Mar;20(2):323-330. doi: 10.5811/westjem.2018.12.41085. Epub 2019 Feb 6. PMID 30881553
- [Background] Kam J, Taylor DM. Obesity significantly increases the difficulty of patient management in the emergency department. Emerg Med Australas. 2010 Aug;22(4):316-23. doi: 10.1111/j.1742-6723.2010.01307.x. PMID 20796008
- [Background] Dargin J, Medzon R. Emergency department management of the airway in obese adults. Ann Emerg Med. 2010 Aug;56(2):95-104. doi: 10.1016/j.annemergmed.2010.03.011. Epub 2010 Apr 3. PMID 20363528
- [Background] Pleskot M, Tilser P, Pidrman V. [The effect of orciprenaline on the heart conduction system]. Bratisl Lek Listy. 1986 Sep;86(3):295-9. No abstract available. Czech. PMID 3756561
- [Background] Peitz GW, Troyer J, Jones AE, Shapiro NI, Nelson RD, Hernandez J, Kline JA. Association of body mass index with increased cost of care and length of stay for emergency department patients with chest pain and dyspnea. Circ Cardiovasc Qual Outcomes. 2014 Mar;7(2):292-8. doi: 10.1161/CIRCOUTCOMES.113.000702. Epub 2014 Mar 4. PMID 24594550
- [Background] Hossain P, Kawar B, El Nahas M. Obesity and diabetes in the developing world--a growing challenge. N Engl J Med. 2007 Jan 18;356(3):213-5. doi: 10.1056/NEJMp068177. No abstract available. PMID 17229948
- [Background] Ding D, Lawson KD, Kolbe-Alexander TL, Finkelstein EA, Katzmarzyk PT, van Mechelen W, Pratt M; Lancet Physical Activity Series 2 Executive Committee. The economic burden of physical inactivity: a global analysis of major non-communicable diseases. Lancet. 2016 Sep 24;388(10051):1311-24. doi: 10.1016/S0140-6736(16)30383-X. Epub 2016 Jul 28. PMID 27475266
- [Background] Ward ZJ, Bleich SN, Long MW, Gortmaker SL. Association of body mass index with health care expenditures in the United States by age and sex. PLoS One. 2021 Mar 24;16(3):e0247307. doi: 10.1371/journal.pone.0247307. eCollection 2021. PMID 33760880
- [Background] Lavie CJ, Ozemek C, Carbone S, Katzmarzyk PT, Blair SN. Sedentary Behavior, Exercise, and Cardiovascular Health. Circ Res. 2019 Mar;124(5):799-815. doi: 10.1161/CIRCRESAHA.118.312669. PMID 30817262
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Hirode G, Wong RJ. Trends in the Prevalence of Metabolic Syndrome in the United States, 2011-2016. JAMA. 2020 Jun 23;323(24):2526-2528. doi: 10.1001/jama.2020.4501. PMID 32573660
- [Background] Stierman B, Afful J, Carroll MD, Chen TC, Davy O, Fink S, Fryar CD, Gu Q, Hales CM, Hughes JP, Ostchega Y, Storandt RJ, Akinbami LJ. National Health and Nutrition Examination Survey 2017-March 2020 Prepandemic Data Files-Development of Files and Prevalence Estimates for Selected Health Outcomes. Natl Health Stat Report. 2021 Jun 14;(158):10.15620/cdc:106273. doi: 10.15620/cdc:106273. PMID 39380201
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Stewart LK, Kline JA. Acceptability of Exercise in Urban Emergency Department Patients With Metabolic Syndrome, Including a Subset With Venous Thromboembolism. J Patient Exp. 2022 Mar 2;9:23743735221083165. doi: 10.1177/23743735221083165. eCollection 2022. PMID 35252559
- [Background] Tang N, Stein J, Hsia RY, Maselli JH, Gonzales R. Trends and characteristics of US emergency department visits, 1997-2007. JAMA. 2010 Aug 11;304(6):664-70. doi: 10.1001/jama.2010.1112. PMID 20699458
- [Background] Boudreaux ED, Cydulka R, Bock B, Borrelli B, Bernstein SL. Conceptual models of health behavior: research in the emergency care settings. Acad Emerg Med. 2009 Nov;16(11):1120-3. doi: 10.1111/j.1553-2712.2009.00543.x. PMID 20053231
- [Background] Boudreaux ED, Bock B, O'Hea E. When an event sparks behavior change: an introduction to the sentinel event method of dynamic model building and its application to emergency medicine. Acad Emerg Med. 2012 Mar;19(3):329-35. doi: 10.1111/j.1553-2712.2012.01291.x. PMID 22435866
- [Background] Montesi L, Moscatiello S, Malavolti M, Marzocchi R, Marchesini G. Physical activity for the prevention and treatment of metabolic disorders. Intern Emerg Med. 2013 Dec;8(8):655-66. doi: 10.1007/s11739-013-0953-7. Epub 2013 May 9. PMID 23657989
- [Background] Sallis R, Franklin B, Joy L, Ross R, Sabgir D, Stone J. Strategies for promoting physical activity in clinical practice. Prog Cardiovasc Dis. 2015 Jan-Feb;57(4):375-86. doi: 10.1016/j.pcad.2014.10.003. Epub 2014 Oct 22. PMID 25459975
- [Background] Petrides J, Collins P, Kowalski A, Sepede J, Vermeulen M. Lifestyle Changes for Disease Prevention. Prim Care. 2019 Mar;46(1):1-12. doi: 10.1016/j.pop.2018.10.003. Epub 2018 Dec 22. PMID 30704651
- [Background] Burgess E, Hassmen P, Pumpa KL. Determinants of adherence to lifestyle intervention in adults with obesity: a systematic review. Clin Obes. 2017 Jun;7(3):123-135. doi: 10.1111/cob.12183. Epub 2017 Mar 15. PMID 28296261
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Background] Eckel RH, Jakicic JM, Ard JD, de Jesus JM, Houston Miller N, Hubbard VS, Lee IM, Lichtenstein AH, Loria CM, Millen BE, Nonas CA, Sacks FM, Smith SC Jr, Svetkey LP, Wadden TA, Yanovski SZ, Kendall KA, Morgan LC, Trisolini MG, Velasco G, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 AHA/ACC guideline on lifestyle management to reduce cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S76-99. doi: 10.1161/01.cir.0000437740.48606.d1. Epub 2013 Nov 12. No abstract available. PMID 24222015
- [Background] Jacobson TA, Maki KC, Orringer CE, Jones PH, Kris-Etherton P, Sikand G, La Forge R, Daniels SR, Wilson DP, Morris PB, Wild RA, Grundy SM, Daviglus M, Ferdinand KC, Vijayaraghavan K, Deedwania PC, Aberg JA, Liao KP, McKenney JM, Ross JL, Braun LT, Ito MK, Bays HE, Brown WV, Underberg JA; NLA Expert Panel. National Lipid Association Recommendations for Patient-Centered Management of Dyslipidemia: Part 2. J Clin Lipidol. 2015 Nov-Dec;9(6 Suppl):S1-122.e1. doi: 10.1016/j.jacl.2015.09.002. Epub 2015 Sep 18. PMID 26699442
- [Background] American Diabetes Association. 10. Cardiovascular Disease and Risk Management: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S111-S134. doi: 10.2337/dc20-S010. PMID 31862753
- [Background] American Diabetes Association. Addendum. 8. Obesity Management for the Treatment of Type 2 Diabetes: Standards of Medical Care in Diabetes-2020. Diabetes Care 2020;43(Suppl. 1):S89-S97. Diabetes Care. 2020 Aug;43(8):1980. doi: 10.2337/dc20-ad08b. Epub 2020 Jun 5. No abstract available. PMID 32503836
- [Background] Nilsson PM, Tuomilehto J, Ryden L. The metabolic syndrome - What is it and how should it be managed? Eur J Prev Cardiol. 2019 Dec;26(2_suppl):33-46. doi: 10.1177/2047487319886404. PMID 31766917
- [Background] Despres JP, Lemieux I. Abdominal obesity and metabolic syndrome. Nature. 2006 Dec 14;444(7121):881-7. doi: 10.1038/nature05488. PMID 17167477
- [Background] Eckel RH, Grundy SM, Zimmet PZ. The metabolic syndrome. Lancet. 2005 Apr 16-22;365(9468):1415-28. doi: 10.1016/S0140-6736(05)66378-7. PMID 15836891
- [Background] Boudreau DM, Malone DC, Raebel MA, Fishman PA, Nichols GA, Feldstein AC, Boscoe AN, Ben-Joseph RH, Magid DJ, Okamoto LJ. Health care utilization and costs by metabolic syndrome risk factors. Metab Syndr Relat Disord. 2009 Aug;7(4):305-14. doi: 10.1089/met.2008.0070. PMID 19558267
- [Background] Stewart LK, Kline JA. Metabolic syndrome increases risk of venous thromboembolism recurrence after acute deep vein thrombosis. Blood Adv. 2020 Jan 14;4(1):127-135. doi: 10.1182/bloodadvances.2019000561. PMID 31917844
- [Background] Stewart LK, Kline JA. Metabolic Syndrome Increases Risk of Venous Thromboembolism Recurrence after Acute Pulmonary Embolism. Ann Am Thorac Soc. 2020 Jul;17(7):821-828. doi: 10.1513/AnnalsATS.201907-518OC. PMID 32187500
- [Background] Stewart LK, Peitz GW, Nordenholz KE, Courtney DM, Kabrhel C, Jones AE, Rondina MT, Diercks DB, Klinger JR, Kline JA. Contribution of fibrinolysis to the physical component summary of the SF-36 after acute submassive pulmonary embolism. J Thromb Thrombolysis. 2015 Aug;40(2):161-6. doi: 10.1007/s11239-014-1155-5. PMID 25433511
- [Background] Vuckovic BA, Cannegieter SC, van Hylckama Vlieg A, Rosendaal FR, Lijfering WM. Recurrent venous thrombosis related to overweight and obesity: results from the MEGA follow-up study. J Thromb Haemost. 2017 Jul;15(7):1430-1435. doi: 10.1111/jth.13710. Epub 2017 May 31. PMID 28439955
- [Background] Eichinger S, Hron G, Bialonczyk C, Hirschl M, Minar E, Wagner O, Heinze G, Kyrle PA. Overweight, obesity, and the risk of recurrent venous thromboembolism. Arch Intern Med. 2008 Aug 11;168(15):1678-83. doi: 10.1001/archinte.168.15.1678. PMID 18695082
- [Background] Borch KH, Braekkan SK, Mathiesen EB, Njolstad I, Wilsgaard T, Stormer J, Hansen JB. Abdominal obesity is essential for the risk of venous thromboembolism in the metabolic syndrome: the Tromso study. J Thromb Haemost. 2009 May;7(5):739-45. doi: 10.1111/j.1538-7836.2008.03234.x. Epub 2008 Nov 24. PMID 19036065
- [Background] Summer R, Walsh K, Medoff BD. Obesity and pulmonary arterial hypertension: Is adiponectin the molecular link between these conditions? Pulm Circ. 2011 Oct-Dec;1(4):440-7. doi: 10.4103/2045-8932.93542. PMID 22530098
- [Background] Molica F, Morel S, Kwak BR, Rohner-Jeanrenaud F, Steffens S. Adipokines at the crossroad between obesity and cardiovascular disease. Thromb Haemost. 2015 Mar;113(3):553-66. doi: 10.1160/TH14-06-0513. Epub 2014 Oct 23. PMID 25338625
- [Background] Steffen LM, Cushman M, Peacock JM, Heckbert SR, Jacobs DR Jr, Rosamond WD, Folsom AR. Metabolic syndrome and risk of venous thromboembolism: Longitudinal Investigation of Thromboembolism Etiology. J Thromb Haemost. 2009 May;7(5):746-51. doi: 10.1111/j.1538-7836.2009.03295.x. Epub 2009 Jan 19. PMID 19175496
- [Background] Ageno W, Dentali F, Grandi AM. New evidence on the potential role of the metabolic syndrome as a risk factor for venous thromboembolism. J Thromb Haemost. 2009 May;7(5):736-8. doi: 10.1111/j.1538-7836.2009.03327.x. Epub 2009 Feb 24. No abstract available. PMID 19245417
- [Background] Ay C, Tengler T, Vormittag R, Simanek R, Dorda W, Vukovich T, Pabinger I. Venous thromboembolism--a manifestation of the metabolic syndrome. Haematologica. 2007 Mar;92(3):374-80. doi: 10.3324/haematol.10828. PMID 17339187
- [Background] Ageno W, Prandoni P, Romualdi E, Ghirarduzzi A, Dentali F, Pesavento R, Crowther M, Venco A. The metabolic syndrome and the risk of venous thrombosis: a case-control study. J Thromb Haemost. 2006 Sep;4(9):1914-8. doi: 10.1111/j.1538-7836.2006.02132.x. Epub 2006 Jul 17. PMID 16848878
- [Background] Samson SL, Garber AJ. Metabolic syndrome. Endocrinol Metab Clin North Am. 2014 Mar;43(1):1-23. doi: 10.1016/j.ecl.2013.09.009. PMID 24582089
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169